CLINICAL TRIAL: NCT03485469
Title: A Prospective Randomized Clinical Trial, in Open-label, Multicenter, Estimating the Impact of the Hypnosis on the Loss of Weight at Patients in Failure of Bariatric Surgery
Brief Title: The Impact of the Hypnosis on the Loss of Weight at Patients in Failure of Bariatric Surgery
Acronym: BARIATHYPNOSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL17_0024; UF 9793 (Other: Montpellier University Hospital)
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Bariatric Surgery
Keywords: Obesity; bariatric surgery; Hypnosis
MeSH Terms: conditions — Obesity | interventions — Hypnosis; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Other): The control group will benefit from a standard care dietary consultation in the service and 9 dietary consultations by phone every 15 days.
  Interventions: Behavioral: Standard Care
- Hypnosis (Other): The experimental group will benefit from a dietary consultation in the service, 9 dietary consultations by telephone every 15 days to which will be associated 7 individual sessions of hypnosis and 3 individual sessions of learning to autohypnosis. A recording containing the induction of a self-hypnosis session will be given to the subject at the end of the 10 sessions, in order to promote the continuation of home-made autohypnosis.
  Interventions: Behavioral: Hypnosis

INTERVENTIONS:
Behavioral: Hypnosis — There ar 10 hypnosis sessions :
  * 1st session of hypnosis : relaxation and orientation towards "emotional cleansing".
  * 2nd session of hypnosis: oriented towards digestion, physical and psychological
  * 3rd session of hypnosis: oriented towards the feeling of security.
  * 4th session of hypnosis: self-esteem oriented.
  * 5th hypnosis session: oriented towards emotional management.
  * 6th hypnosis session: oriented towards self-confidence.
  * 7th hypnosis session: oriented towards the completion of the projects.
  * 8th, 9th and 10th sessions: concern the learning of self-hypnosis and autonomy. A USB key containing the induction of a session of autohypnosis will be given to the subject to promote the continuation of home-made auto-hypnosis.
  Arms: Hypnosis
Behavioral: Standard Care — The dietary advice given during these dietary consultations is part of the standard care adapted to patients who have undergone bariatric surgery while increasing the frequency of consultations (Fractionation of meals, Volume of meals, Taking meals, Drinks, Food diversity)
  Arms: Usual Care

SUMMARY:
The therapeutic problem of obesity is weight control, a major difficulty, involving a significant change in eating behavior. A number of studies show that there are many factors of resistance to weight loss whether they are physiological, genetic, environmental pressure related, or psychological and behavioral. For some patients, the surgical approach seems the best alternative. Indeed, bariatric surgery is an effective therapeutic weapon in patients with morbid obesity. However, it has been shown that approximately 25% of patients are failing at two years of this surgery (Reinhold's index). Some of the failed subjects may benefit from surgical revision. As for the others, no intervention is currently proposed to them. Studies have shown that the psychological profile of patients who are candidates for bariatric surgery is predominantly impulsive, very anxious with a tendency to depression. The stress level of these patients would be important, and they would have low self-esteem. This study hypothesize that, in these patients, the establishment of hypnotherapeutic management associated with the usual dietary monitoring could modify eating habits thus promoting weight loss and an improvement in self-esteem , stress and anxiety compared to dietary monitoring alone.

DETAILED DESCRIPTION:
he therapeutic problem of obesity is weight control, a major difficulty, involving a significant change in eating behavior. A number of studies show that there are many factors of resistance to weight loss whether they are physiological, genetic, environmental pressure related, or psychological and behavioral. For some patients, the surgical approach seems the best alternative. Indeed, bariatric surgery is an effective therapeutic weapon in patients with morbid obesity. However, it has been shown that approximately 25% of patients are failing at two years of this surgery (Reinhold's index). Some of the failed subjects may benefit from surgical revision. As for the others, no intervention is currently proposed to them. Studies have shown that the psychological profile of patients who are candidates for bariatric surgery is predominantly impulsive, very anxious with a tendency to depression. The stress level of these patients would be important, and they would have low self-esteem. This study hypothesize that, in these patients, the establishment of hypnotherapeutic management associated with the usual dietary monitoring could modify eating habits thus promoting weight loss and an improvement in self-esteem , stress and anxiety compared to dietary monitoring alone.

There are still no studies assessing the impact of hypnotherapeutic management and self-hypnosis on the weight curve, self-esteem, stress, anxiety, or the quality of life of patients Obese in failure of bariatric surgery.

It is an Interventional, prospective, multi-center, controlled, randomized, open-label study with 2 parallel arms, evaluating the efficacy of hypnotherapeutic management in patients with bariatric surgery failure, compared to dietary monitoring alone.

Number of visits: 13 visits are planned: 1 visit of inclusion, a visit ensuring the first dietary follow-up, 9 hypnosis sessions (for the experimental group), two visits dedicated to the collection of the judgment criteria. Each patient is followed for 12 months.

The estimated duration of recruitment is 18 months.

ELIGIBILITY:
Inclusion criteria:

* Obese patient (BMI = 30 kg / m ²)
* 18 - 65 years ( inclusive borders)
* Patient in failure of bariatric surgery and in which no surgical resumption can be proposed (in view of Reinhold's classification, the failure will be considered as a loss of overweight lower than 50 % in two years further to a bariatric surgery).
* Informed consent
* Patient in measure to realize all the visits and to follow the procedures of the study - Subject affiliated to a social security system

Exclusion criteria:

* Pregnancy current or planned during the duration of the study, pregnant or breast-feeding women
* Craniopharyngioma or any other evolutionary malignant pathology, or chronic illness in decompensation phase
* Strong probability of not compliance to the protocol or drop-out
* Psychiatric pathology of dissociated type (schizophrenia; psychosis, bipolarity …)
* Sensory (hearing, visual) or cognitive deficits susceptible to hinder the progress of the sessions.
* Incapacity to understand the nature and the purpose of the study and\or communication difficulties with the investigator
* Patient having already benefited from a coverage by hypnotherapy for loss of weight
* Taken by treatment having an impact on the loss of weight (corticoid, antithyroid …)
* Major protected by the law or considered vulnerable (under guardianship)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in weight in 5 months | 5 months
  Patient weight (in kg) measurement will be performed on the same scale by staff who are unaware of the patient's randomization group.

SECONDARY OUTCOMES:
Change in weight in 12 months | 12 months
  Patient weight (in kg) measurement will be performed on the same scale by staff who are unaware of the patient's randomization group.
Self-esteem | 12 months
  It will be evaluated by the scale of "Rosenberg's Self Esteem Scale" (1965) validated in French. It represents an assessment of the overall self-esteem that the person can have of herself. The scale includes 10 statements measured on a scale of 1 to 4.
Evolution of Quality of life | 12 months
  it will be evaluated by the variation of the scores obtained in the self-questionnaire EQVOD (Echelle de Qualité de Vie, Obésité et Diététique) of O. Ziegler et al (2005). It's a specific quality of life questionnaire for obese people.
Anxiety and depressive state | 12 months
  It will be evaluated by the Hospital Anxiety and Depression Scale - HAD (Sigmond et al, 1983). It is a self-administered 14-item questionnaire that assesses the current level of depressive and anxious symptomatology by eliminating somatic depressions that may skew assessments.
Feeding behavior | 12 months
  It will be evaluated by the TFEQ-R21 (Three-Factor Eating Questionnaire) self-questionnaire (Cappelleri et al, 2009).
  TFEQ has been validated in the general population and has been used in many studies. It explores three components of eating behavior: cognitive restriction, uncontrolled eating, and emotional eating.
Patients' satisfaction with their care | 12 months
  It will be evaluated the Likert scales of the self-satisfaction questionnaire. It is composed of 5 Likert scales coded from 1 to 5 which will be analyzed separately

CONTACTS AND LOCATIONS:
Overall Officials: David NOCCA, PU-PH, Principal Investigator — University Hospital, Montpellier
Locations (5):
- France (5):
  - CHR Saint Pierre - maladies métaboliques, La Réunion
  - Cécile GODEL, Montpellier
  - Orléans University Hospital, Orléans
  - Reims University Hospital, Reims
  - Toulouse University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No